CLINICAL TRIAL: NCT05136729
Title: The Effects of Face-to-Face vs Online Self-Natural Posture Exercise Programs on Chronic Low Back Pain
Brief Title: The Effects of Self-Natural Posture Exercise Programs on Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Billings Clinic (Other)
Collaborators: SNPE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21.011; SNPE 09.02.2021 (Other: Billings Clinic)
Record Dates: First submitted 2021-11-16; First posted 2021-11-29 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Chronic Low-back Pain
Keywords: therapeutic; rehabilitation; stabilization; behavioral
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled trial (RCT) design with a wait-list control group
Who Masked: Outcomes Assessor
Masking Description: Care providers and investigators are blinded to outcome assessment. The de-identified data will be provided to the biostatistician for analysis. Analyzed data will be submitted to the PI for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face Self-Natural Posture Exercise training (Experimental): Off-line training
  Interventions: Behavioral: Self-Natural Posture Exercise training
- Online Self-Natural Posture Exercise training (Active Comparator): Virtual training
  This group as a wait-list control group will receive online SNPE intervention after serving as an untreated comparison group.
  Interventions: Behavioral: Self-Natural Posture Exercise training

INTERVENTIONS:
Behavioral: Self-Natural Posture Exercise training — SNPE training will be provided face-to-face or online by certified instructors. The SNPE exercise training involves the use of special belts to align and stabilize posture and joints. Up to 4 belts can be used, placed around the hips, around the thighs, below the knees, and above the ankles. Myofascial release is part of the training, which is self-performed with SNPE equipment.
  Other Names: SNPE training

SUMMARY:
Low back pain is a major health problem across the United States, with socio-economic burden, major cause of disability, and poor quality of life. One such non-pharmacologic treatment is Self-Natural Posture Exercise (SNPE), a series of exercise programs developed in conjunction with orthodontic bracing principles. Belts are worn around the hips (pelvic correction belt) and legs (right posture belt) to assist with self-directed exercise and posture correction. A typical SNPE program has eight different movements, targeting the entire axial skeleton. The exercises can be practiced anywhere and are widely applicable to patients as exercises are low- to moderate-intensity flexibility-based muscle strength training. There are several studies from Korea examining the efficacy of SNPE; however, there are few English language studies and there are no studies from outside the country of South Korea. As such, there is little data the generalizability of SNPE, the degree of cultural acceptance in other countries, and the all-important adherence to the home exercise program. The present study proposes to be the first study outside of South Korea to examine the effects of SNPE on chronic low back patients.

DETAILED DESCRIPTION:
The present study seeks to repeat the previously described positive clinical impact of SNPE in a new population, examine rates of adherence, and compare the effects of face-to-face versus online courses.

Specific Aims:

1. Aim 1: Investigate the adherence to an SNPE program in American adults to explore the generalizability of existing Korean data.
2. Aim 2: Assess the effects of a 12-week face-to-face vs online SNPE program on back pain. We hypothesize that the face-to-face group will show greater pain reduction and improvements in body posture and quality of life compared to the control group after phase 1.
3. Aim 3: Compare adherence to and effects of face-to-face vs online 12-week SNPE programs.
4. Aim 4: Investigate the adherence to and effects of face-to-face vs online 12-week SNPE programs at a follow-up of 12 weeks.

A single-blind randomized controlled trial (RCT) design with a wait-list control group will be used to evaluate the effect of SNPE for back pain reduction. The control group will receive online SNPE intervention after serving as an untreated comparison group. The wait-list control group serves two purposes. First, it provides an untreated comparison for the face-to-face group to determine if the intervention had an effect. By serving as a comparison group, researchers are able to isolate the independent variable and look at the impact it had. Second, it allows the wait-listed participants an opportunity to obtain the intervention at a later date.

Recruitment:

Flyers, Billings Clinic employee emails, and social media will be used to recruit participants. Recruitment messages will include relevant information about the study, benefits, and inclusion criteria as well as a link to a study-specific website recapitulating this information (https://xppizim.wixsite.com/snpestudy). When patients contact the investigators, any questions will be answered. If the patient chooses to go forward, the ODI Questionnaire and Self-reported Data Form will be collected online (www.surveymonkey.com). Data will be reviewed for eligibility, and if appropriate, participant will be sent the information contained on the consent form to review; the actual signed form will be collected at time of their 1st assessment prior to the collection of data.

After being assessed by a physiatrist, eligible participants will be invited to participate in the study. All participants will have an equal chance of being randomly assigned (using a random number table from Microsoft Excel to produce random numbers).

Analyses:

All data will be exported from www.surveymonkey.com and analyzed using the Statistical Package for Social Sciences (SPSS) application. Descriptive statistics will be used to summarize demographic variables. To investigate adherence mentioned in Aim 1 and 4, frequencies and percentages will be analyzed for categorical variables and mean, standard deviation, quartiles, and ranges for continuous variables. For Aim 2 and 3, all outcome measures will be compared between groups (Assessment 1 will be considered the baseline for face-to-face (FTF) and Assessment 2 will be the baseline for online (ONL)), will be analyzed using an analysis of covariance (ANCOVA) via the General Linear Model (GLM). Age and gender will be controlled as covariates. If there is a significant difference using ANCOVA, we will follow up with post hoc testing.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-65 yr
* Body mass index (BMI): 18.5-34.9
* Low back disability index: 16-50% (moderate low back pain)
* Internet access with mobile device or desktop sufficient for video streaming
* No plan to have back pain treatment (opioid medication, physical therapy, and/or other procedures) in the next 12 months

Exclusion Criteria:

* Have had spine or pelvic orthopedic or neurologic surgery
* Have history or evidence of functionally significant musculoskeletal deformity
* Have history or evidence of functionally significant balance dysfunction
* Have a significant medical (e.g., cardiac or pulmonary) condition
* Are or plan to become pregnant
* Not currently receiving manual or physical interventions for low back pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline low back disability (measured by ODI) at week 0, 12, 24, and 36 | Specific metric will be gathered at outset of study and then after a 12 week intervention. It will be gathered again 12 weeks further out (24 weeks from outset). It will be gathered again 12 weeks further out (36 weeks).
  Questionnaire: Oswestry Disability Index (ODI). Patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. Questionnaire examines perceived level of disability in 10 everyday activities of daily living.
Mean change from baseline pain (measured by VAS) at week 0, 12, 24, and 36 | Specific metric will be gathered at outset of study and then after a 12 week intervention. It will be gathered again 12 weeks further out (24 weeks from outset). It will be gathered again 12 weeks further out (36 weeks).
  The Visual Analog Scale (VAS). The pain VAS is a unidimensional measure of pain intensity. Patients rate their subjective pain on a scale from 0 to 10, with zero being no pain and 10 being the worst pain imaginable.
Mean change from baseline quality of life (measured by SF-36) at week 0, 12, 24, and 36 | Specific metric will be gathered at outset of study and then after a 12 week intervention. It will be gathered again 12 weeks further out (24 weeks from outset). It will be gathered again 12 weeks further out (36 weeks).
  The 36-Item Short Form Survey (SF-36). It is a 36 question self reported measure of health and crosses 8 domains including but not limited to physical, mental, and social health.
Mean change from baseline muscle tone (measured by Myoton Pro device, in Hz) at week 0, 12, 24, and 36 | Specific metric will be gathered at outset of study and then after a 12 week intervention. It will be gathered again 12 weeks further out (24 weeks from outset). It will be gathered again 12 weeks further out (36 weeks).
  Muscle tone is a biomechanical characteristic of a muscle and is measured as the muscle's natural vibration in a stable state without voluntary muscle contraction. This is expressed in frequency (㎐), and the higher the value, the higher the muscle tension. Muscle tone will be measured using a non-invasive muscle tone meter developed for objective quantification of the mechanical properties of muscles.
Mean change from baseline pain (measured by FPX25 device, in kg/cm^2) at week 0, 12, 24, and 36 | Specific metric will be gathered at outset of study and then after a 12 week intervention. It will be gathered again 12 weeks further out (24 weeks from outset). It will be gathered again 12 weeks further out (36 weeks).
  Pain by site will be evaluated by pressure pain threshold (PPT). PPT is defined as the minimum force applied which induces pain and is an indicator of sensitivity to pain. The examiner will place a flat circular (1㎠) probe attached to the digital pressure gauge vertically on the measured muscle and pressure will be gradually applied. When the examiner releases the probe, the pressure at the time of removal appears on the screen in units of kg/cm^2.
Mean change from baseline body alignment (measured by dartfish software, in angular degrees) at week 0, 12, 24, and 36 | Specific metric will be gathered at outset of study and then after a 12 week intervention. It will be gathered again 12 weeks further out (24 weeks from outset). It will be gathered again 12 weeks further out (36 weeks).
  Posture alignment will be evaluated by photographing standing posture of study participants from the front and side and images will be analyzed using Dartfish software.

CONTACTS AND LOCATIONS:
Overall Officials: Younsun Son, PhD, Principal Investigator
Locations (1):
- Billings Clinic, Billings, Montana, United States

IPD SHARING:
Plan to Share IPD: No